CLINICAL TRIAL: NCT00269412
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess The Efficacy and Safety of Three Different Doses (275, 550 AND 1100 MG) of Rifaximin Administered BID For Either Two or Four Weeks in The Treatment of Patients With Diarrhea-Associated Irritable Bowel Syndrome
Brief Title: Study to Assess the Efficacy and Safety of Rifaximin Administered BID in the Treatment of Patients With Diarrhea-Associated Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RFIB2001
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin

INTERVENTIONS:
Drug: Rifaximin

SUMMARY:
This is placebo-controlled study of three rifaximin doses in patients with DIBS. Subjects will be randomized to receive daily doses of placebo BID, rifaximin 275 mg BID, rifaximin 550 mg BID, or 1100 mg BID for 14 days. These four groups will subsequently receive an additional two weeks of placebo for a total of 4 weeks of treatment. A fifth group of subjects will receive rifaximin 550 mg BID for a period of 28 days. Subjects who successfully respond to treatment at the end of the 28-day Treatment Phase will be followed in a Post-treatment Phase that includes study visits during Weeks 6, 8, 12 and 16. Subjects who relapse during the Post-treatment Phase will be discontinued from the study.

DETAILED DESCRIPTION:
While IBS is one of the most common chronic medical conditions the etiology of IBS is unknown. Although not a life-threatening illness, IBS is considered to be a serious condition that has a substantial impact on a subject's day-to-day function. IBS is characterized by abdominal pain and altered bowel habits, including diarrhea, constipation, or alternating diarrhea and constipation. Symptoms are typically intermittent but may be continuous.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18 years of age or older.
2. Irritable bowel syndrome confirmed by the Rome II Criteria
3. Lower endoscopic examination that demonstrates normal colonic anatomy

Exclusion Criteria:

1. Subject has exclusively constipation-predominant IBS (CIBS) that is characterized by < 3 bowel movements/week or hard and lumpy stools.
2. Subject has alternating IBS, but is currently presenting with constipation associated IBS symptoms.
3. Subject has had adequate control of their DIBS and their symptom of bloating the week preceding the screening visit or at the time of randomization. Bloating includes the following symptoms: abdominal fullness, bloating, gas, or swelling.
4. Subjects has a positive stool culture for O & P (ovum and parasite) and/or Clostridium difficile
5. Subject has failed to record 2 negative weekly global assessments during the past 10 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate the efficacy of a 14-day course of oral rifaximin at 550 mg BID versus placebo in providing adequate relief from Diarrhea-associated IBS (DIBS) symptoms.

SECONDARY OUTCOMES:
To evaluate the dose-response relationship of placebo administered for 28 days and rifaximin administered at 275 mg BID, 550 mg BID, or 1100 mg BID for 14 days;
to evaluate the efficacy of 550 mg BID for 4 weeks to determine if there are any differences when treatment is extended for an additional 2-week period when compared to a similar dosing regimen for 2 weeks;
to evaluate the durability of response over a 12-week Post-treatment Phase in subjects with DIBS who achieved a response during the acute Treatment Phase of the study.

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Premeire Pharmaceutical Research, Tempe, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Lovelace Scientific Resources, Irvine, California
  - West Gastroenterology Medical Group, Los Angeles, California
  - Beverly Hills Gastroenterology, Los Angeles, California
  - Medical Associates Research Group, San Diego, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Litchfield County Gastroenterology Associates, LLC, Torrington, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - University Clinical Research, DeLand, Florida
  - Research Consultants Group, Hialeah, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Shafran Gastroenterology, Winter Park, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Rockford Gastroenterology, Rockford, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Gastrointestinal Clinic of Quad Citites, Davenport, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Digestive Disorders Associates, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Maryland Clinical Trials, Severna Park, Maryland
  - Capital Gastroenterology Consultants, PA, Silver Springs, Maryland
  - Coastal Research Associates, Braintree, Massachusetts
  - Henry Ford Hospital, Chesterfield, Michigan
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Gastroenterology and Hepatology, Kansas City, Missouri
  - Center for Digestive & Liver Diseases, Inc., Mexico, Missouri
  - Specialist in Gastroenterology, St Louis, Missouri
  - Gastroenterology Specialities, Lincoln, Nebraska
  - Long Island Clinical Research, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Vital re:Search, Greensboro, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Bethany Medical Center, High Point, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Digestive Health Network, Cincinnati, Ohio
  - GI & Liver Diseases Consultants, Dayton, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Digestive Health Specialists, PA, Oklahoma City, Oklahoma
  - West Hills Gastroenterology Associates, PC, Portland, Oregon
  - Columbia Gastroenterology Associates, Columbia, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Regional Research Institute, Jackson, Tennessee
  - Holston Valley Physicians, Kingsport, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - Advanced Research Institute, Ogden, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Internal Medicine Associates, Danville, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - North Pacific Clinical Research, Redmond, Washington
  - Spokane Digestive Disease Center, Spokane, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Schoenfeld P, Pimentel M, Chang L, Lembo A, Chey WD, Yu J, Paterson C, Bortey E, Forbes WP. Safety and tolerability of rifaximin for the treatment of irritable bowel syndrome without constipation: a pooled analysis of randomised, double-blind, placebo-controlled trials. Aliment Pharmacol Ther. 2014 May;39(10):1161-8. doi: 10.1111/apt.12735. Epub 2014 Apr 3. PMID 24697851